CLINICAL TRIAL: NCT05388721
Title: Correlation Between Environmental Pollution and Gestational Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: Environment2022
Record Dates: First submitted 2022-05-15; First posted 2022-05-24 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GDM group: Pregnant women with positive OGTT results at 24-28 gestational weeks
  Interventions: Other: Clinical data and specimen collection
- Control group: Pregnant women with negative OGTT results at 24-28 gestational weeks, and had baseline data that matched those in the GDM group
  Interventions: Other: Clinical data and specimen collection

INTERVENTIONS:
Other: Clinical data and specimen collection — Questionnaire survey and clinical data was conducted when pregnant women were enrolled in the first trimester, and blood and urine were collected. Furthermore, we will follow up the pregnant women until delivery, blood and urine were collected during the third trimester (after 28 weeks), and clinical information was collected.
  Umbilical cord blood and placental tissue will be collected if possible.

SUMMARY:
Gestational diabetes mellitus (GDM) refers to the abnormal glucose metabolism index of pregnant women during pregnancy. At present, about 15% of pregnant women will develop GDM in the second and third trimester, which seriously affects the health of the pregnant woman and the fetus. However, the etiology of GDM remains unclear. Various pollutants in the environment may have a potential impact on pregnant women and fetuses. For example, previous studies have shown that exposure to atmospheric pollutants nitric oxide and organochlorine pesticides are associated with GDM. At present, we plan to further investigate the correlation between environmental pollutants and GDM.

ELIGIBILITY:
Inclusion Criteria:

* Plan to complete OGTT and give birth in the research center
* First trimester
* Singleton pregnancy
* Without diabetes before pregnancy

Exclusion Criteria:

* Have diseases that affect metabolic function or even threaten the life of the mother and fetus before pregnancy, such as diabetes, hypertension, heart disease, liver and kidney diseases, thyroid diseases with drug, autoimmune diseases, malignant tumors, AIDS, etc.
* Fetus has a known deformity or genetic defects
* Incomplete clinical data
* Assisted reproductive

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This project intends to recruit pregnant women who go to the research center for routine prenatal examination and OGTT screening.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Environmental contaminants 1 | First trimester (9-14 gestational weeks)
  The concentrations of environmental pollutants, such as organochlorine pesticides, polychlorinated biphenyls, polycyclic aromatic hydrocarbons, polybrominated diphenyl ethers and metallic elements, in serum and urine were analyzed by gas chromatochromatograms and mass spectrometry (GC-MS/MS). Specimens were collected during the first trimester and tested when classified in the GDM or control group
Environmental contaminants 2 | Third trimester (after 28 gestational weeks)
  The concentrations of environmental pollutants, such as organochlorine pesticides, polychlorinated biphenyls, polycyclic aromatic hydrocarbons, polybrominated diphenyl ethers and metallic elements, in serum and urine were analyzed by gas chromatochromatograms and mass spectrometry (GC-MS/MS). Specimens were collected during the third trimester.

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Hospital School Of Medicine Zhejiang University, Hangzhou, Zhejiang, China